CLINICAL TRIAL: NCT03169842
Title: Accuracy of Cyst Fluid Glucose for the On-site Diagnosis of Mucinous Pancreatic Cysts
Brief Title: Cyst Fluid Glucose for On-site Diagnosis of Mucinous Pancreatic Cysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016.227.C
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cyst fluid glucose (Experimental): Single arm- cyst fluid glucose will be measured from pancreatic cyst fluid aspirate
  Interventions: Device: pancreatic cyst fluid glucose analysis using a bedside glucometer

INTERVENTIONS:
Device: pancreatic cyst fluid glucose analysis using a bedside glucometer — Small amount of pancreatic cyst fluid will be analyzed for glucose level using a bedside glucometer from EUS-FNA procedures.

SUMMARY:
This study evaluates the utility of using cyst fluid glucose levels to diagnose mucinous pancreatic cysts during endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) procedures.

DETAILED DESCRIPTION:
Mucinous pancreatic cysts are considered pre-cancerous. The standard evaluation of pancreatic cysts usually includes endoscopic ultrasound-guided fine needle aspiration (EUS-FNA). The cyst fluid sample from EUS-FNA is routinely sent for lab analysis (carcinoembryonic antigen-CEA) and cytology assessment. The diagnosis of a mucinous cyst is usually based on those results.

For study participants undergoing EUS-FNA, a small portion of the cyst fluid will be analyzed for glucose levels using a bedside glucometer in addition to the routine analyses. A low cyst fluid glucose level may correlate with a diagnosis of a mucinous cyst. The primary aim of this study will be to determine if a low cyst fluid glucose level correlates with standard laboratory cyst fluid analysis (CEA) in establishing a diagnosis of a mucinous pancreatic cyst.

Secondary aims of this study will be: (1) comparing the accuracy of cyst fluid glucose to CEA level among subjects with a proven diagnosis of a mucinous cyst (based on surgery or cytopathology findings), and (2) determining the optimal cyst fluid glucose level that correlates to a proven diagnosis of a mucinous cyst (based on subjects who undergo surgery or have a diagnosis based on cytopathology).

ELIGIBILITY:
Inclusion Criteria:

* All adults undergoing standard-of-care EUS-FNA procedures for the evaluation of pancreatic cysts are eligible to participate
* Minimum of 1mL of cyst fluid must be aspirated in order to be enrolled in the study

Exclusion Criteria:

* Inability to perform pancreatic cyst fluid sampling
* <1mL of cyst fluid is aspirated during EUS-FNA

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Cyst fluid glucose level | immediate, point-of-care measurement at time of EUS-FNA of pancreatic cyst fluid
  concentration of cyst fluid glucose based on measurement with bedside glucometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No